CLINICAL TRIAL: NCT04644692
Title: Positive Diagnosis of Heart Failure With Preserved LVEF by Exercise Pulmonary Ultrasound.
Brief Title: Effort-Lung Ultra Sound
Acronym: E-LUS
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Mathieu ECHIVARD, Praticien hospitalier, Central Hospital, Nancy, France
Other Study IDs: 2020PI156
Record Dates: First submitted 2020-11-12; First posted 2020-11-25 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: patients with heart failure with preserved ejection fraction
  Interventions: Other: Lung ultrasound
- Control Group:Never diagnosed with either preserved or altered ejection fraction heart failure.: Non dyspnoeic patients with no history of Heart failure.
  Interventions: Other: Lung ultrasound

INTERVENTIONS:
Other: Lung ultrasound — A lung ultrasound before and at the end of the stress test.

SUMMARY:
The E-LUS study is a prospective, non randomised, monocenter case-control study.

The main objective is to evaluate the association of exercise lung ultrasound data acquired during a stress test on a bicycle ergometer with the diagnosis of heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
Secondary objectives:

1. To assess the diagnostic performance of exercise lung ultrasound for the diagnosis of HFpEF.
2. To identify the value of the B-lines score on exercise maximizing the sensitivity and specificity for the diagnosis of HFpEF.
3. To evaluate the relationship of the delta of B-lines scores between rest and exercise with the diagnosis of HFpEF.
4. To assess the diagnostic performance of the delta of B-lines between rest and exercise for the diagnosis of HFpEF.
5. To identify the score of the delta of B-lines value between rest and exercise maximizing sensitivity and specificity for the diagnosis of HFpEF.
6. To evaluate the relationship between the resting value of the B-lines scores with the diagnosis of HFpEF.
7. To assess the diagnostic performance of the resting lung ultrasound for the diagnosis of HFpEF.
8. To identify the value of the B-lines score at rest maximizing the sensitivity and specificity for the diagnosis of HFpEF.
9. To evaluate the correlation between the B-line score measured at rest and exercise and the dyspnoea score measured at rest, during exercise, and during the recovery phase.
10. To assess the correlation of the delta of B-lines scores between rest and exercise and the dyspnoea score measured at rest, during exercise and during the recovery phase.

ELIGIBILITY:
Inclusion Criteria (Control group) :

* Patients 65 years of age and older scheduled for a stress test.
* Never diagnosed with either preserved or altered ejection fraction heart failure
* Non-dyspneic (New York Heart Association class I)

Inclusion Criteria (Case group) :

* Patients 65 years of age and older scheduled for a stress test.
* Patients already diagnosed with HFpEF following hospitalization for heart failure (LVEF>50%)

Exclusion Criteria:

* Patients who are opposed to participate to the research project / the use of their data,
* Pulmonary or pleural pathology preventing reliable acquisition of lung ultrasound images (e.g. pulmonary fibrosis, diffuse interstitial lung disease or lung cancer)
* Patients with a history of thoracic surgery
* Patients under legal protection measures (guardianship, curator, judicial safeguard),
* Pregnant women, parturient women or nursing mothers,
* Patients who are unable to express consent,
* Persons deprived of their liberty by a judicial or administrative decision,
* Persons subject to psychiatric care,
* Patients discharged from hospital for a worsening heart failure hospitalization for less than 15 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged 65 years and older scheduled for a stress test.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
The exercise B-lines score measured by the 8-point method. | Within 2 minutes after the end of the stress test
  This score can have a value from 0 to 80, each anterior thoracic measurement point being rated from 0 to 10. A higher value indicate a higher level of pulmonary congestion. The measurement will be taken at the end of the stress test, in the first 2 minutes of recovery

SECONDARY OUTCOMES:
The diagnosis of HFpEF, as defined by a history of hospitalization for acute heart failure with preserved Left Ventricular Ejection Fraction (LVEF). | Within 10 minutes prior the start of the stress test
  For secondary objectives 1, 2, 4, 5, 7 and 8, the endpoint will be the diagnosis of HFpEF, as defined by a history of hospitalization for acute heart failure with preserved LVEF.
2. The delta of B-lines scores during exercise measured by the 8-point method between rest and the end of the exercise | Between Within 10 minutes prior the start of the stress test and 2 minutes after the end of the stress test
  Regarding secondary objective 6, the judgment criterion will be the score of B-lines at rest measured by the 8-point method within 10 minutes prior the start of the stress test. This score can have a value from 0 to 80, each anterior thoracic measurement point being rated from 0 to 10. A higher value indicate a higher level of pulmonary congestion.
The B-lines score at rest measured by the 8-point method | Within 10 minutes prior the start of the stress test
The modified Borg dyspnea score at rest, during exercise and during recovery. | Within 10 minutes prior the start of the stress test, at the peak of exercise and 3 minutes after the end of the stress test
  For secondary objectives 9 and 10, the endpoint will be the modified Borg dyspnea score at rest, during exercise and during recovery. This scale is ranging from 0 to 10, 10 indicating a maximal level of dyspnea.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France